CLINICAL TRIAL: NCT05951530
Title: The Impact of App-based Cognitive Training on Post-stroke Upper Extremity Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0207
Record Dates: First submitted 2023-05-09; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Stroke
Keywords: stroke, sub-acute stroke, cognitive impairment
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy (Active Comparator): This group will receive conventional upper extremity rehabilitation including active and active assisted ROMs and upper extremity stretches for 30 minutes, three to five times a week for 6 weeks.
  Interventions: Other: traditional physical therapy
- The impact of app-based cognitive training (Experimental): The experimental group received mobile-app-based cognitive training (PEAK) along with conventional upper extremity rehabilitation.
  Interventions: Other: mobile app-based cognitive training

INTERVENTIONS:
Other: traditional physical therapy — this group received conventional upper extremity active ROMs and stretches for 30 minutes three to five times a week for 6 weeks without using the app-based cognitive training.
  Arms: Traditional physical therapy
Other: mobile app-based cognitive training — This group received mobile app-based cognitive training of 30minutes session three to five times a week for 6 weeks which includes a few activities such as the memory, coordination and alertness along with conventional UE exercises for 15 minutes three to five times a week for 6 weeks.
  Arms: The impact of app-based cognitive training

SUMMARY:
To find out the impact of app-based cognitive training on upper extremity function in patients with sub-acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45-70 years.
* Both male and female gender.
* Patients of sub-acute stroke patients with impaired upper extremity function
* Stroke patients suffering from mild to moderate cognitive impairment.
* Patients with the ability to fulfill and comprehend commands

Exclusion Criteria:

* Patients of neurodegenerative diseases like Parkinson's, multiple sclerosis etc.
* Patients suffering from any severe psychological disorder.
* Patients with severe contracture due to orthopedic disease of the shoulder, elbow, and wrist joints

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
upper extremity function | 4th week
  Fugl-Meyer Assessment-Upper Extremity (FMA-UE) The FMA-UE is a condition-specific outcome that applies to hemiparesis of the upper limb in stroke conditions. The FMA motor assessments for the upper (maximum score 66 points)
Trail Making Test | 4th week
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It has two parts, in which the subject is instructed to connect a set of 25 dots as quickly as possible while maintaining accuracy. Scoring is based on time taken to complete the test (e.g. 35 seconds yielding a score of 35) with lower scores being better. Different norms are available that allow comparison with age-matched groups

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- sir Ganga Ram Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feigin VL, Krishnamurthi RV, Parmar P, Norrving B, Mensah GA, Bennett DA, Barker-Collo S, Moran AE, Sacco RL, Truelsen T, Davis S, Pandian JD, Naghavi M, Forouzanfar MH, Nguyen G, Johnson CO, Vos T, Meretoja A, Murray CJ, Roth GA; GBD 2013 Writing Group; GBD 2013 Stroke Panel Experts Group. Update on the Global Burden of Ischemic and Hemorrhagic Stroke in 1990-2013: The GBD 2013 Study. Neuroepidemiology. 2015;45(3):161-76. doi: 10.1159/000441085. Epub 2015 Oct 28. PMID 26505981
- [Background] Kim YD, Jung YH, Saposnik G. Traditional Risk Factors for Stroke in East Asia. J Stroke. 2016 Sep;18(3):273-285. doi: 10.5853/jos.2016.00885. Epub 2016 Sep 30. PMID 27733028
- [Background] Nomani AZ, Nabi S, Badshah M, Ahmed S. Review of acute ischaemic stroke in Pakistan: progress in management and future perspectives. Stroke Vasc Neurol. 2017 Feb 24;2(1):30-39. doi: 10.1136/svn-2016-000041. eCollection 2017 Mar. PMID 28959488
- [Background] Langhorne P, Legg L. Evidence behind stroke rehabilitation. J Neurol Neurosurg Psychiatry. 2003 Dec;74 Suppl 4(Suppl 4):iv18-iv21. doi: 10.1136/jnnp.74.suppl_4.iv18. No abstract available. PMID 14645462
- [Background] Levin MF, Kleim JA, Wolf SL. What do motor "recovery" and "compensation" mean in patients following stroke? Neurorehabil Neural Repair. 2009 May;23(4):313-9. doi: 10.1177/1545968308328727. Epub 2008 Dec 31. PMID 19118128
- [Background] Engfeldt B, Hultenby K, Muller M. Ultrastructure of hyaline cartilage. I. A comparative study of cartilage from different species and locations, using cryofixation, freeze-substitution and low-temperature embedding techniques. Acta Pathol Microbiol Immunol Scand A. 1986 Sep;94(5):313-23. PMID 3532690
- [Background] Tang EY, Amiesimaka O, Harrison SL, Green E, Price C, Robinson L, Siervo M, Stephan BC. Longitudinal Effect of Stroke on Cognition: A Systematic Review. J Am Heart Assoc. 2018 Jan 15;7(2):e006443. doi: 10.1161/JAHA.117.006443. PMID 29335318
- [Background] Pinter D, Enzinger C, Gattringer T, Eppinger S, Niederkorn K, Horner S, Fandler S, Kneihsl M, Krenn K, Bachmaier G, Fazekas F. Prevalence and short-term changes of cognitive dysfunction in young ischaemic stroke patients. Eur J Neurol. 2019 May;26(5):727-732. doi: 10.1111/ene.13879. Epub 2019 Jan 9. PMID 30489673
- [Background] McDonald MW, Black SE, Copland DA, Corbett D, Dijkhuizen RM, Farr TD, Jeffers MS, Kalaria RN, Karayanidis F, Leff AP, Nithianantharajah J, Pendlebury S, Quinn TJ, Clarkson AN, O'Sullivan MJ. Cognition in stroke rehabilitation and recovery research: Consensus-based core recommendations from the second Stroke Recovery and Rehabilitation Roundtable. Int J Stroke. 2019 Oct;14(8):774-782. doi: 10.1177/1747493019873600. Epub 2019 Sep 12. PMID 31514685
- [Background] Wiley E, Khattab S, Tang A. Examining the effect of virtual reality therapy on cognition post-stroke: a systematic review and meta-analysis. Disabil Rehabil Assist Technol. 2022 Jan;17(1):50-60. doi: 10.1080/17483107.2020.1755376. Epub 2020 May 2. PMID 32363955
- [Background] Fruhwirth V, Enzinger C, Fandler-Hofler S, Kneihsl M, Eppinger S, Ropele S, Schmidt R, Gattringer T, Pinter D. Baseline white matter hyperintensities affect the course of cognitive function after small vessel disease-related stroke: a prospective observational study. Eur J Neurol. 2021 Feb;28(2):401-410. doi: 10.1111/ene.14593. Epub 2020 Nov 12. PMID 33065757